CLINICAL TRIAL: NCT06874972
Title: Effect of Music Therapy on the Quality of Recovery in Patients Undergoing Laparoscopic Cholecystectomy Under General Anesthesia, at the National Referral Hospital, Bhutan: a Randomized Controlled Trial
Brief Title: Effect of Music Therapy on the Quality of Recovery
Acronym: MTonR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ministry of Health, Bhutan (Other Government)
Responsible Party: Principal Investigator, Yeshey Dorjey, Effect of music therapy on the quality of recovery in patients undergoing laparoscopic cholecystectomy under general anesthesia, at the national referral hospital, Bhutan: a randomized controlled trial, Ministry of Health, Bhutan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Music for recovery
Record Dates: First submitted 2025-02-14; First posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Music Therapy; Music Therapy for Pain and Sedation; Postoperative Period; Perioperative Period; Visual Analog Scale
Keywords: music therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Music group) (Experimental): Music is played to the study group (music group)
  Interventions: Device: Music played
- Control group (no music played) (No Intervention): No music is played in the control group

INTERVENTIONS:
Device: Music played — Music is played in the study group, and no music is played in the control group.
  Arms: Study group (Music group)

SUMMARY:
Background:

The use of music in operations is increasing due to its painless, safe, inexpensive, and the potential to improve patient outcomes.

Objective:

We aimed to evaluate the effects of music therapy on the quality of awakening and recovery of patients who underwent elective laparoscopic cholecystectomy under general anesthesia, and to compare the perioperative pain and anxiety related to surgery.

Methods:

This double-blinded randomized clinical trial was conducted at the National Referral Hospital, Bhutan from 1st November 2022 to 31st October 2023. Those patients who underwent laparoscopic cholecystectomy under general anesthesia were included in the clinical trial. Web-based simple randomization was performed, and all those patients with even numbers were allocated to the study group and odd numbers in the control group. During the perioperative period, music was played using headphones in the study group, and empty headphone was placed in the control group. Hemodynamic parameters, quality of awakening (measured using the Riker sedation-agitation scale), and recovery (measured using a 40-item questionnaire, QoR-40) were recorded using a questionnaire developed for the study. Perioperative anxiety and pain were compared between the study group using a Visual analog scale (VAS).

DETAILED DESCRIPTION:
INTRODUCTION Music is a structured combination of sound with recognizable melody and rhythm, that is pleasant or exciting to listen to. Music causes body and mind relaxation, improves mood, reduces stress, and improves memory.

Music modulates the release of neurotransmitters in the brain. Musical stimuli increase extracellular levels of dopamine and serotonin and have pleasant effects on the body and mind.

Due to its pleasant effects on the body and mind, music has been used as a therapy in the medical field. Music therapy is found to significantly decrease pain, improve emotional distress from pain, reduce anesthetic agents and opioid use, and improve heart rate, blood pressure, and saturation during surgical procedures.

Music is usually played in the operating theatres. Music has an impact on the operating teams. Few surgeons and operating teams have regarded music as a distraction to their task, however, the positive impact of music on the surgical performance of the surgeons and the operating teams and the surgical outcomes was reported significantly more compared to the negative impact.

Patients prefer to listen to different music depending on their likes during the perioperative period. Music is found to have a positive impact on patients waiting for surgery by reducing stress, anxiety, and depression.

Despite music having multiple positive impacts on patients and the operating teams, there is limited evidence on the effect of music on the postoperative recovery of patients from anesthesia and surgery.

Therefore, this study aimed to evaluate the impact of music on the quality of awakening and recovery of patients who underwent laparoscopic cholecystectomy under general anesthesia at the national referral hospital, in Bhutan.

MATERIALS AND METHODS This double-blinded randomized control trial compared the effects of music on the quality of arousal, quality of recovery, and patient satisfaction between the music group and control group. It was conducted at the Jigme Dorji Wangchuk (JDW) National Referral Hospital, Bhutan, over a period of one year from 1st November 2022 to 31st October 2023. All those patients who underwent laparoscopic cholecystectomy under general anesthesia at JDW National Referral Hospital during the study period were eligible for the study.

All patients undergoing laparoscopic cholecystectomy under general anesthesia with American Society of Anesthesiologists (ASA) Grade I and II were included.

Patients with ASA III or more, patients with hearing or cognitive impairment, patients with ear infections (acute or chronic suppurative otitis media) and with recent ear surgery, patients on long-term steroid therapy, those with drug or alcohol abuse history, those unable to cooperate (due to dementia and mental retardation) were excluded.

This study is presented following the Consolidated Standards of Reporting Trials (CONSORT)[10] guidelines. An ethical clearance was obtained from the Institutional Review Board of Khesar Gyalpo University of Medical Sciences of Bhutan (KGUMSB) [11] with Ref No: IRB/Approval/PN/2022-018/ 445, dated 10th November 2022.

Before the commencement of the study, the investigators trained the doctors and nurses on the study procedure. Anesthesia personnel and obstetricians were informed to perform TAP for the intervention group and to infiltrate along the CS wound in the comparator group. The nurses of the PACU, and maternity ward were trained on the study procedure of collecting the data on pain scores using VAS, recording the opioids used during the postoperative period, and postoperative complications.

The investigators approached those pregnant mothers posted for elective CS during the pre-operative period. Pregnant women were counseled and informed about the trial 1 day before the scheduled CS. Information on the multimodal treatment for postoperative pain including administration of local anesthetic in the transversus abdominis plane under ultrasound guidance and or infiltration along the cesarean section wound was shared with them. Written informed consent was obtained from the mothers who agreed to participate in the study. Those mothers fulfilling the inclusion criteria were recruited for the study. After recruitment, pregnant mothers were briefed and familiarised with the visual analog scale (VAS) for pain scores.

Simple randomization was done through computerized randomization. This was a double-blinded randomized trial where the researchers and the study participants did not know which intervention they received.

Study procedure:

After the recruitment of the patients, the demographic variables (age, gender, and BMI) and the ASA classifications were collected in a research questionnaire. The patients were taken for the scheduled operation for laparoscopic cholecystectomy under general anesthesia. The starting time of anesthesia was recorded as the time of induction of anesthesia. General anesthesia was administered following standard protocol of the institutes for all the patients. After administering the anesthesia, a skin incision was performed which was recorded as the starting time of surgery. Patients in both groups had standard monitoring during the surgical procedure with electrocardiogram, blood pressure, and pulse oximetry. Heart rate, systolic blood pressure, diastolic blood pressure, and mean arterial pressure, were recorded after induction and every 5 minutes of anesthesia and immediately after extubation. All hemodynamic parameter measurements were accomplished with MINDRAY anesthesia equipment, which was validated according to the hospital's biomedical engineering standard operating procedure.

The completion of the surgical procedure was recorded as the end of skin closure, and the extubation of the endotracheal tube was recorded as the end of anesthesia time.

After extubation, patients were taken to the post-anesthetic care unit (PACU) for recovery, where routine vitals were monitored. Once the patient had fully recovered from anesthesia, they were shifted to the surgical ward.

Intervention:

After the induction of anesthesia headphone labeled with number 1 was put on to patients belonging to group 1 and headphone labeled as 2 was put on to the patients in group 2. The headphones were linked to a music player and covered using the operation theatre drapes for further blinding. Patients allocated in group 1 were attached to headphone 1, and the music player was activated (contained song), and in group 2, headphone 2 was attached and activated the music player (contained no song).

In headphone 1, the intensity of the music sound was set at a level of 60 decibels with the help of an audiometer from the Audiology Unit. The headphones employed for this study were JBL T450BT on-ear wireless headphones. They were lightweight and comfortable which had minimum impact on the ears. The leather ear cushions made them easy to apply and clean. The sound produced was well-balanced with good bass and treble. It offered up to 11 hours of playback time on a single charge. The music player was an Apple iPod, where sounds were adjusted to certain frequencies based on hearing needs. The extensive features of the iPod, quality, and comparably low price made it a good choice for this trial. In group 1, relaxing classical instrumental music was played in repeat mode. Music was played after the induction, throughout the surgery until the end of the surgery (completion of skin closure), and extubation, and fully awakened and recovered from the anesthesia.

Study tools:

A pretested interviewer-administered questionnaire was used for the collection of the data. Demographic variables were collected. All the patients were assessed for the quality of arousal and pain score at PACU. The quality of arousal was assessed using the Riker sedation-agitation scale [13] and the pain score was rated using a visual analog score (VAS) [14] at the PACU. The Riker sedation-agitation scale has scores ranging from 1 to 7 (score 1- unarousable, score 2- very sedated, score 3- sedated, score 4- calm and cooperative, score 5- agitated, score 6- very agitated, and score 7- dangerous agitated). Postoperative pain was rated using a VAS, which has a score of 0 indicating no pain, to a score of 10 indicating unbearable pain.

After 24 hours of operation in the surgical ward, the quality of recovery and patient satisfaction were assessed using a standard 40-item questionnaire (QoR-40) which consisted of five dimensions. This QoR-40 is a pre-tested and validated questionnaire to evaluate the quality of recovery after surgery.[15] These five dimensions are emotional state, physical comfort, psychological support, physical independence, and pain, which consist of 9, 12, 7, 5, and 7 responses respectively. Individual responses in each domain scored from 1 very poor to 5 excellent. The emotional state domain has a minimum score of 9 to a maximum of 45 scores; physical comfort has a minimum of 12 and a maximum of 60 scores; psychological support has a minimum of 7 and a maximum of 35 scores; physical independence has a minimum of 5 and maximum 25 scores and pain domain has minimum 7 and a maximum of 35 scores. The overall or the Global QoR-40 has a minimum of 40 and a maximum score of 200. More scores recorded in the domains are considered better quality recovery and more satisfied patients during the postoperative period.

Follow-up:

Patients were transferred to PACU after the laparoscopic cholecystectomy and monitored for vitals. The quality of arousal was assessed using the Riker sedation-agitation scale, and the pain score was rated using a visual analog score (VAS) at the PACU. Patients were transferred to the surgical ward once hemodynamically stable. After 24 hours of operation in the surgical ward, the quality of recovery and patient satisfaction were assessed using a standard 40-item questionnaire (QoR-40) as detailed above in the study tool.

Sample size:

The sample size was calculated using the G*Power version 3.1.97. The sample size obtained was 78, and with a drop rate of 5%, the total sample size (n) was 84, which was equally divided into two groups, the music group (n=) and the control group (n=42).

Data management:

Daily data were cross-checked by the principal investigator for completeness.

Data analysis:

Data were double-entered and validated using EpiData (version 3.1 for entry and version 2.2.2.183 for analysis, EpiData Association, Odense, Denmark).

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing laparoscopic cholecystectomy under general anesthesia
* Patients with American Society of Anesthesiologists (ASA) Grade I and II

Exclusion Criteria:

* Patients with ASA III or more
* Patients with hearing or cognitive impairment
* Patients with ear infections (acute or chronic suppurative otitis media) and with recent ear surgery
* Patients on long-term steroid therapy
* Patients with drug or alcohol abuse history
* Patients who are unable to cooperate (due to dementia and mental retardation)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Quality of awakening | 12 months
  To compare the quality of awakening from surgery and anesthesia between study and control group using Riker sedation-agitation scale
Quality of recovery from surgery and anesthesia | 12 months
  To compare qaulity of recovery from surgery and anesthesia between study and control group using Riker sedation-agitation scale

SECONDARY OUTCOMES:
Postoperative pain score | 12 months
  To compare postoperative pain score between study and control group using Visual analog scale (VAS)

CONTACTS AND LOCATIONS:
Overall Officials: Yeshey Dorjey, Principal Investigator — Phuentsholing General Hospital
Locations (1):
- Phuentsholing Hospital, Phuentsholing, Bhutan